CLINICAL TRIAL: NCT01697566
Title: An Endometrial Cancer Chemoprevention Study of Metformin Versus No Treatment in Women With a Body Mass Index (BMI) >/= 30 kg.m2 and Hyperinsulinemia
Brief Title: An Endometrial Cancer Chemoprevention Study of Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-0739; 5P50CA098258 (NIH); NCI-2013-00834 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Gynecology
Keywords: Gynecology; Endometrial Cancer Chemoprevention; Obese; Body Mass Index (BMI) >/= 35 kg.m2; Post-menopausal; Hyperinsulinemia; Metformin; Placebo; Sugar pill; Lifestyle intervention; Diet; Exercise
MeSH Terms: conditions — Obesity; Hyperinsulinism; Motor Activity | interventions — Metformin; Sugars; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Metformin (Experimental): Participants gradually increase the dose of metformin by mouth as listed below:
  Week 1: One capsule each day Week 2: One capsule 2 times each day Week 3: One capsule 3 times each day Week 4: Two capsules 2 times each day
  After week 4, participant continues to take 2 capsules of metformin 2 times each day.
  Each capsule is 425 mg.
  Interventions: Drug: Metformin; Procedure: Endometrial Biopsy; Behavioral: Questionnaires
- Placebo + Lifestyle Intervention (Experimental): Placebo taken by mouth twice daily for 4, 30 day cycles. Lifestyle intervention consists of 16 in-person sessions offered over a 4 month period.
  Interventions: Other: Placebo; Procedure: Endometrial Biopsy; Behavioral: Lifestyle Intervention; Behavioral: Questionnaires
- Metformin + Lifestyle Intervention (Experimental): Participants gradually increase the dose of metformin by mouth as listed below:
  Week 1: One capsule each day Week 2: One capsule 2 times each day Week 3: One capsule 3 times each day Week 4: Two capsules 2 times each day
  After week 4, participant continues to take 2 capsules of metformin 2 times each day.
  Each capsule is 425 mg.
  Lifestyle intervention consists of 16 in-person sessions offered over a 4 month period.
  Interventions: Drug: Metformin; Procedure: Endometrial Biopsy; Behavioral: Lifestyle Intervention; Behavioral: Questionnaires
- Placebo (Placebo Comparator): Placebo taken by mouth twice daily for 4, 30 day cycles.
  Interventions: Other: Placebo; Procedure: Endometrial Biopsy; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Metformin — Participants gradually increase the dose of metformin by mouth as listed below:
  Week 1: One capsule each day Week 2: One capsule 2 times each day Week 3: One capsule 3 times each day Week 4: Two capsules 2 times each day
  After week 4, participant continues to take 2 capsules of metformin 2 times each day.
  Each capsule is 425 mg.
  Arms: Metformin; Metformin + Lifestyle Intervention
Other: Placebo — Placebo taken by mouth twice daily for 4, 30 day cycles.
  Other Names: sugar pill
  Arms: Placebo; Placebo + Lifestyle Intervention
Procedure: Endometrial Biopsy — Endometrial biopsies obtained at baseline and after 4 months.
Behavioral: Lifestyle Intervention — Lifestyle intervention consists of 16 in-person sessions offered over a 4 month period.
  Arms: Metformin + Lifestyle Intervention; Placebo + Lifestyle Intervention
Behavioral: Questionnaires — Completion of questionnaires about diet and exercise at baseline, during treatment and at end of study. Questionnaires take about 30-40 minutes to complete.
  Other Names: surveys

SUMMARY:
The goal of this clinical research study is to learn about the effects of metformin and/or a program called "lifestyle intervention" on the endometrium (inner lining of the uterus) in post-menopausal women who are also obese (both are risk factors for endometrial cancer). Researchers also want to learn how insulin levels will be affected by metformin, diet and/or exercise.

Metformin is designed to treat both diabetes and insulin resistance. Insulin resistance is a condition in which the body makes insulin but does not use it properly. It is often referred to as "pre-diabetes". Many people with insulin resistance have high levels of both sugar and insulin in their blood at the same time, which have been reported in patients with endometrial cancer.

In this study, metformin will be compared to a placebo. A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

Lifestyle intervention is made up of a series of in-person sessions where you meet with a coach to discuss strategies for losing weight and ways to increase physical activity. It also consists of materials designed to help you lose weight and will offer opportunities for supervised exercise.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the roll of dice) to 1 of 4 study groups:

* Metformin only.
* Placebo and lifestyle intervention.
* Metformin and lifestyle intervention.
* Placebo only.

Neither you nor the study staff will know if you are receiving metformin or placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

In the first month you will gradually increase the dose of metformin/placebo by mouth as listed below:

* Week 1: One capsule each day
* Week 2: One capsule 2 times each day
* Week 3: One capsule 3 times each day
* Week 4: Two capsules 2 times each day

After week 4, you will continue to take 2 capsules of metformin/placebo 2 times each day.

If you are receiving the lifestyle intervention, you will have 16 lifestyle intervention sessions over 4 months. At each of these sessions, you will discuss methods for managing your weight. You will receive print materials and worksheets, measuring utensils, and a food scale. You will be instructed how to use each of these materials and how often to use them during the study. You will also be provided with opportunities for supervised exercise (such as group exercise class and group walks).

If you are traveling during a scheduled session, it can be performed over the telephone. Each call should last about 30 minutes, during which you will discuss the same goals and information that you would discuss in the in-person sessions.

Study Visits:

Before you can begin receiving the study drug/placebo:

* At the second screening visit , you will have a dual energy x-ray absorptiometry (DEXA) scan to measure your body composition. The scan requires you to lie still on a table for about 8-10 minutes while a low-energy x-ray takes an image that allows the study staff to get an image of your body fat density.
* You will be given an accelerometer (a small, portable device that measures your physical activity) and be taught how to use it at the first Screening Visit. You will wear the accelerometer at all times while you are awake for 7 days. At the second Screening Visit, you will return the accelerometer at an intervention session. If you are not able to return it at the second visit then you will mail it back to the study staff in a pre-paid envelope. You will receive the accelerometer again at Month 4 and wear it for another 7 days.
* You will receive a study diary in which you will record any and all exercise you perform each day while you are on study. It should take about 5 minutes to complete each time.
* You will complete questionnaires about diet and exercise. These questionnaires should take about 30-40 minutes to complete.
* You will also be taught to complete a questionnaire on the internet to record the food you eat in a 24 hour period. You will do this 3 times over a 2 week period. The first time, you will complete it at the clinic. The study staff will call and remind you to complete the questionnaire the other 2 times. Each time you complete this questionnaire, it should take about 40 minutes.

At Month 1, all participants will return for a study visit. The following tests and procedures will be performed:

* Blood (about 2 teaspoons) will be drawn for routine tests. If this blood draw shows that your liver or kidney function is abnormal, you will need to return for an additional blood °draw at Month 2.
* If you are having symptoms that you would describe as moderate or worse, you will have a non-pelvic physical exam including measurement of your vital signs and any unreported symptoms you may be having.

At each month, you will be asked about any symptom(s) that you may have to learn if it is related to the study. If you are called, this phone call should last about 5 minutes. If you are asked in a in-person visit, the visit can last up to an hour.

Length of Study:

You will receive the study drug/placebo and/or lifestyle intervention for up to 4 months. You will be taken off study if you have intolerable side effects or if you develop endometrial cancer or hyperplasia during the study. Your participation in the study will be over after the end-of-study visit.

Post-Treatment Visit:

At the end of the 4th month, you will have a post-treatment visit. You will repeat all procedures performed in the first and second visit:

* Your height, weight, waist, and hip circumference will be measured.
* You will have a DEXA scan.
* You will complete the questionnaires about food, diet, and exercise.
* You will be given a questionnaire about your satisfaction (based on the intervention) to complete and return at this visit. This questionnaire will take up to an hour to complete.
* You will have an endometrial biopsy.
* Blood (about 8 tablespoons) will be drawn for routine tests and for biomarker testing. You will have to fast (not eat or drink anything except water) for 12 hours before this blood draw.
* You will complete the questionnaire on the internet to record the food you eat in a 24 hour period. You will do this 3 times over a 2 week period. The first time, you will complete it at the clinic. The study staff will call and remind you to complete the questionnaire the other 2 times. Each time you complete this questionnaire, it should take about 40 minutes.

Follow-Up:

About 1 year after the screening visits (+/- 1 month), the following tests and procedures will be performed:

* Your height, weight, waist, and hip circumference will be measured.
* You will have a DEXA scan.
* Blood (about 8 tablespoons) will be drawn for routine tests and for biomarker testing. °You will have to fast (not eat or drink anything except water) for 12 hours before this blood draw.
* You will wear the accelerometer for 7 days.
* You will complete questionnaires about food, diet, and exercise.
* You will complete the questionnaire on the internet to record the food you eat in a 24 hour period. You will do this 3 times over a 2 week period. The first time, you will complete it at the clinic. The study staff will call and remind you to complete the questionnaire the other 2 times. Each time you complete this questionnaire, it should take about 40 minutes.

This is an investigational study. Metformin is FDA approved and commercially available for the treatment of diabetes and insulin resistance.

Up to 100 patients will take part in this study. All will be enrolled at MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. For this study, only women will be enrolled.
2. Body Mass Index (BMI) > or = 30 kg/m2
3. Not frankly diabetic, as measured by a fasting blood glucose </=126 mg/dL.
4. Demonstrate hyperinsulinemia with a QUICK I value </= 0.357.
5. Age >/= 50 and </= 65
6. Zubrod Performance Scale 0-1
7. Hemoglobin >/= 10 g/dl
8. TSH 0.27 - 4.20 µlU/mL
9. Menopause as defined as no menses for 1 year and/or FSH >/= 25.8 mIU/ml
10. Must be able to read, write, and speak English.
11. Must have a Primary Care Provider (PCP).

Exclusion Criteria:

1. Prior hysterectomy or endometrial ablation
2. ALT >/r = 2.0x Upper Limit of Normal (ULN)
3. Serum creatinine > /= 1.4 mg/dl
4. Triglycerides (fasting) >/ = 400
5. Known inability to participate in the ongoing appointments for the four months of the study and scheduled follow-up tests.
6. Significant medical or psychiatric history which would make the participant a poor protocol candidate, in the opinion of the principal investigator, for any aspect of study participation including metformin, unsupervised exercise program or dietary behavior change.
7. Participant reported history of congestive heart failure
8. Prior treatment with Metformin
9. Currently being treated for diabetes or meeting criteria for new diagnosis of diabetes.
10. Known allergy to Metformin or other biguanide (Proguanil).
11. Use of Aromatase Inhibitors, GNRH-agonists i.e.Lupron, Zoladex within the last 6 months
12. Use of SERMS (selective estrogen receptor modulators) in the past 6 months, including Tamoxifen and Raloxifene
13. Hormone replacement therapy within the last 6 months
14. Women who have been treated with chemotherapy for prior malignant disease or currently have an untreated malignancy other than non-melanoma skin cancer
15. Patients who have had prior radiation to the pelvis

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-05-30 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen H. Lu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from May 2013 until May 2016 and all recruitments were done in a medical clinic setting.
Groups:
- Metformin + Lifestyle: Metformin 1700 mg daily along with lifestyle intervention program
- Metformin + No Lifestyle: Metformin 1700 mg daily with no lifestyle intervention program
- Placebo + Lifestyle: Placebo given daily along with lifestyle intervention program
- Placebo + No Lifestyle: Placebo given daily with no lifestyle intervention program
Period: Overall Study
Arm/Group | Metformin + Lifestyle | Metformin + No Lifestyle | Placebo + Lifestyle | Placebo + No Lifestyle
Started | 7 | 7 | 7 | 8
Completed | 7 | 7 | 5 | 7
Not Completed | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Final biopsy not obtained | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin + Lifestyle | Metformin + No Lifestyle | Placebo + Lifestyle | Placebo + No Lifestyle | Total
Number analyzed (Participants) | 7 | 7 | 7 | 8 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 7 | 8 | 29
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 56.3 [50 to 61] | 56 [50 to 65] | 57 [53 to 61] | 59.8 [54 to 65] | 57.4 [50 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 7 | 8 | 29
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 4 | 4 | 2 | 4 | 14
  Unknown or Not Reported | 3 | 2 | 3 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 2 | 4 | 12
  White | 2 | 5 | 4 | 2 | 13
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 7 | 8 | 29

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Participant Body Weight in Pounds (Lbs)
Description: This study will use a 2 x 2 randomized design with all 100 post- menopausal subjects being randomized to metformin, placebo, placebo and intensive lifestyle intervention, or metformin and intensive lifestyle intervention. Treatments will last 4 months. Participants will be assessed at baseline and end of treatment with endometrial sampling to see if there are changes in the biomarkers.
Time Frame: Visit 2 (1 week), 4 months, and 1 year
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Metformin + Lifestyle | Metformin + No Lifestyle | Placebo + Lifestyle | Placebo + No Lifestyle
Number analyzed (Participants) | 7 | 7 | 5 | 7
lbs
  Weight Visit 2 | 108.57 (22.51) | 99.3 (15.36) | 101.64 (13.44) | 94.1 (12.89)
  Weight Month 4 | 101.19 (22.47) | 96.39 (15.36) | 97.98 (16.46) | 94.37 (13.46)
  Weight Year 1 | 102.08 (35.32) | 95.93 (12.63) | 93.25 (8.15) | 94.96 (13.68)
Statistical Analysis 1: Comparison: Metformin + Lifestyle vs Placebo + Lifestyle; Body Weight; Test type: Superiority; p = 0.006, t-test, 2 sided
Statistical Analysis 2: Comparison: Metformin + Lifestyle vs Placebo + Lifestyle; Fat Mass; Test type: Superiority; p < 0.001, t-test, 2 sided

2. Primary Outcome: To Evaluate the Percentage of Ki-67 Positive Cells
Description: The Q-PCR analyses will be performed in the Quantitative Genomics Core Facility at the University of Texas Medical School at Houston.
  Over the last 3 years we have used several techniques including differential display, microchip array screening, and real-time quantitative PCR to find such genes. The tools we have developed are directly applicable to the investigation of surrogate endpoint biomarkers (SEBs). Identification of appropriate biomarkers is essential for this study.
Time Frame: Visit 2 (1 week), 4 months, and 1 year
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Metformin + Lifestyle | Metformin + No Lifestyle | Placebo + Lifestyle | Placebo + No Lifestyle
Number analyzed (Participants) | 7 | 7 | 5 | 7
percentage of cells
  Visit 2 | 8.78 (8.29) | 7.95 (5.13) | 9.23 (3.96) | 4.73 (1.39)
  Month 4 | 6.73 (4.17) | 4.98 (3.94) | 4.17 (2.37) | 9.1 (5.96)

3. Secondary Outcome: BMI
Time Frame: Visit 2 (1 week), 4 months, and 1 year
Measure: Mean (Standard Deviation); unit: weight (kg) / height (m)2
Arm/Group | Metformin + Lifestyle | Metformin + No Lifestyle | Placebo + Lifestyle | Placebo + No Lifestyle
Number analyzed (Participants) | 7 | 7 | 5 | 7
weight (kg) / height (m)2
  BMI Visit 2 | 45.25 (9.36) | 38.17 (5.18) | 39.49 (4.71) | 35.29 (4)
  BMI Month 4 | 39.83 (7.82) | 37.34 (4.78) | 37.83 (5.53) | 35.31 (4.16)
  BMI Year 1 | 41.13 (13.45) | 37.18 (4.41) | 36 (2.3) | 35.54 (4.23)
Statistical Analysis 1: Comparison: Metformin + Lifestyle; Test type: Superiority; p = 0.019, t-test, 2 sided

4. Secondary Outcome: Weight Loss
Time Frame: Visit 2 (1 week), 4 months, and 1 year
Measure: Mean (Standard Deviation); unit: percentage of weight loss
Arm/Group | Metformin + Lifestyle | Metformin + No Lifestyle | Placebo + Lifestyle | Placebo + No Lifestyle
Number analyzed (Participants) | 7 | 7 | 5 | 7
percentage of weight loss
  Weight Loss (Month 4 - Visit 2)/Visit 2 | -7.10 (5.22) | -2.95 (2.34) | -3.88 (5.11) | 0.25 (1.61)
  Weight Loss (Year 1 - Visit 2)/Visit 2 | -5.49 (13.51) | -3.09 (3.45) | -3.37 (4.92) | 0.83 (0.95)

ADVERSE EVENTS:
Time Frame: An average of 36 months
Description: NCI CTCAE version 4.03
Arm/Group | Metformin + Lifestyle | Metformin + No Lifestyle | Placebo + Lifestyle | Placebo + No Lifestyle
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 4/7 | 6/7 | 4/7 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin + Lifestyle (N=7) | Metformin + No Lifestyle (N=7) | Placebo + Lifestyle (N=7) | Placebo + No Lifestyle (N=8)
Flatulence (Gastrointestinal disorders) | 2 (7) | 4 (12) | 2 (6) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 5 (11) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (4) | 4 (8) | 3 (4) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (5) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (8) | 0 (0) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-05-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT01697566/Prot_SAP_000.pdf